CLINICAL TRIAL: NCT06788158
Title: Clinical Effects of the Intralesional Application of Incobotulinum Toxin vs Corticosteroid in Patients With Plantar Fascitis
Brief Title: Clinical Effects of Incobotulinum Toxin vs Corticosteroid in Plantar Fascitis
Acronym: fascitis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Carlos Pech Arguelles, Head of the botulinum toxin application clinic at HGR No.1 IMSS-Yucatán, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-3201-115
Record Dates: First submitted 2025-01-03; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Plantar Fasciitis of Both Feet; Pain; Function
Keywords: botulinum toxin; plantar fasciitis; corticosteroid; pain; foot functionality
MeSH Terms: conditions — Pain; Fasciitis, Plantar | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- incobotulinum toxin + rehabilitation (Experimental): will be administered 2 ampoules (200 IU) of Incobotulinum toxin , injectable solution presentation 100 IU ampoule with powder diluted in 1 ml of 0.9% saline solution in a single application at 4 points, in addition to a therapeutic exercise program in the teaching service to later do it at home that will be done daily for 4 months (cryotherapy for 15 minutes on the plantar fascia, active mobilizations of the ankle and foot for 5 minutes, stretching exercises for the triceps surae and plantar fascia for 20 seconds, 3 repetitions, strengthening of intrinsic muscles of the foot).
  Interventions: Drug: Incobotulinum Toxin A
- glucocorticoid + rehabilitation (Active Comparator): 2 ml of dexamethasone will be administered in an 8 mg/2 ml ampoule diluted in 2 ml of lidocaine injectable solution in a 50 ml bottle (20 mg/ml) in a single application at 1 point, in addition to a therapeutic exercise program in the teaching service to later do it at home that will be done daily for 4 months (cryotherapy for 15 minutes on the plantar fascia, active mobilizations of the ankle and foot for 5 minutes, stretching exercises for the triceps surae and plantar fascia for 20 seconds, 3 repetitions, strengthening of intrinsic muscles of the foot).
  Interventions: Drug: Glucocorticoid

INTERVENTIONS:
Drug: Incobotulinum Toxin A — will be administered 2 ampoules (200 IU) of Incobotulinum toxin , injectable solution presentation 100 IU ampoule with powder diluted in 1 ml of 0.9% saline solution in a single application at 4 points, in addition to a therapeutic exercise program in the teaching service to later do it at home that will be done daily for 4 months (cryotherapy for 15 minutes on the plantar fascia, active mobilizations of the ankle and foot for 5 minutes, stretching exercises for the triceps surae and plantar fascia for 20 seconds, 3 repetitions, strengthening of intrinsic muscles of the foot).
  Arms: incobotulinum toxin + rehabilitation
Drug: Glucocorticoid — Program in which 2 ml of dexamethasone will be administered in an 8 mg/2 ml ampoule diluted in 2 ml of lidocaine injectable solution in a 50 ml bottle (20 mg/ml) in a single application at 1 point, in addition to a therapeutic exercise program in the teaching service to later do it at home that will be done daily for 4 months (cryotherapy for 15 minutes on the plantar fascia, active mobilizations of the ankle and foot for 5 minutes, stretching exercises for the triceps surae and plantar fascia for 20 seconds, 3 repetitions, strengthening of intrinsic muscles of the foot).
  Arms: glucocorticoid + rehabilitation

SUMMARY:
Objectives: To evaluate the clinical effects of intralesional application of incobotulinum toxin vs corticosteroid in patients with plantar fasciitis .

Material and methods: Prospective, experimental, randomized, controlled clinical study; the population will be recruited in the outpatient clinic of the rehabilitation service meeting the inclusion criteria, two randomized study groups will be formed: GROUP A: Patients who accept intralesional infiltration with incobotulinum toxin . GROUP B: Patients who accept intralesional infiltration with dexamethasone.

Both groups will be assessed before application, at 1 month, at 2 and 4 months post intervention. The visual analogue scale (VAS), the American Orthopaedic Foot and Ankle Society (AOFAS) scale and the Foot and Ankle Disability Index (FADI) will be used to assess pain, foot functionality, functional disability index in activities of daily living, in physical activity and measurement of the dorsiflexion arch in 2 visits at the beginning of diagnosis and at 4 months, collecting the variables and establishing a hypothesis analysis to accept or discard normality criteria of the same with tendency and its significance in relation to p <0.05 to establish contrast of the results with parametric or non-parametric variables according to whether or not the hypothesis of normality is discarded.

DETAILED DESCRIPTION:
The investigators want to compare the effects on pain, ankle and foot functionality, as well as activities of daily living; of the application of incobotulinum toxin vs corticosteroid in people suffering from plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Any sex.
3. Diagnosis of plantar fasciitis (pain in the medial plantar calcaneal tubercle which gives rise to the site of plantar fascial insertion into the heel bone and/or pain along the path of its three bands) made by a physician specializing in Physical Medicine and Rehabilitation.
4. Voluntary acceptance of participation in the study.
5. Patients entitled to the Mexican Social Security Institute.

Exclusion Criteria:

1. Diagnosis of ankylosing spondylitis.
2. Pregnant women.
3. Previous infiltration treatment with any medication or substance applied to the plantar fascia or gastrocnemius muscles in the last six months.
4. Anticoagulant treatment.
5. History of local infection in the plantar fascia in the last three months.
6. Allergic to lidocaine, incobotulinum toxin or dexamethasone.
7. Patients not entitled to the Mexican Social Security Institute.
8. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | Initially, 4, 8 and 16 weeks.
  zero is equivalent to no pain and 10 indicates the worst possible pain
Clinical Functional Status of the Ankle and Foot | Initially, 4, 8 and 16 weeks.
  Result of the total summative score of the American Foot and Ankle Society Scale, Excellent=90-100, Good =80-89, Medium=70-79, Poor=<70.
Index of Functional Disability of the Foot and Ankle in Activities of Daily Living | Initially, 4, 8 and 16 weeks.
  Result of the total summative score of the Ankle disability index scale. Absence of disability or pain = 100 Mild=80-99 Moderate=50-79 Severe:1-49 Maximum disability level = 0
Index of Functional Disability of the Foot and Ankle in Sports Activities | Initially, 4, 8 and 16 weeks.
  Result of the total summative score of the ankle disability index scale. Absence of disability or pain = 100 Mild=80-99 Moderate=50-79 Severe:1-49 Maximum disability level = 0

SECONDARY OUTCOMES:
Mobility Arc | Initially and 16 weeks.
  Range of motion (degree of travel) or total angular/axial displacement allowed at ankle joint, dosiflexion degrees at the time of data collection, will be expressed in the results by mobility range groups according to the American Academy of Orthopedic Surgeons AAOS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Regional No.1 "Lic. Ignacio García Téllez" IMSS, Calle 41 101, Fénix, 97155 Mérida, Yuc., Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dressler D. Clinical Pharmacology of Botulinum Toxin Drugs. Handb Exp Pharmacol. 2021;263:93-106. doi: 10.1007/164_2019_273. PMID 32886157
- [Background] Dressler D, Johnson EA. Botulinum toxin therapy: past, present and future developments. J Neural Transm (Vienna). 2022 Jun;129(5-6):829-833. doi: 10.1007/s00702-022-02494-5. Epub 2022 Apr 9. PMID 35396965
- [Background] Camargo CP, Xia J, Costa CS, Gemperli R, Tatini MD, Bulsara MK, Riera R. Botulinum toxin type A for facial wrinkles. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD011301. doi: 10.1002/14651858.CD011301.pub2. PMID 34224576
- [Background] Choudhury S, Baker MR, Chatterjee S, Kumar H. Botulinum Toxin: An Update on Pharmacology and Newer Products in Development. Toxins (Basel). 2021 Jan 14;13(1):58. doi: 10.3390/toxins13010058. PMID 33466571
- [Background] Chou AC, Ng SY, Koo KO. Endoscopic Plantar Fasciotomy Improves Early Postoperative Results: A Retrospective Comparison of Outcomes After Endoscopic Versus Open Plantar Fasciotomy. J Foot Ankle Surg. 2016 Jan-Feb;55(1):9-15. doi: 10.1053/j.jfas.2015.02.005. Epub 2015 May 23. PMID 26007627
- [Background] Li Z, Xia C, Yu A, Qi B. Ultrasound- versus palpation-guided injection of corticosteroid for plantar fasciitis: a meta-analysis. PLoS One. 2014 Mar 21;9(3):e92671. doi: 10.1371/journal.pone.0092671. eCollection 2014. PMID 24658102
- [Background] Elizondo-Rodriguez J, Araujo-Lopez Y, Moreno-Gonzalez JA, Cardenas-Estrada E, Mendoza-Lemus O, Acosta-Olivo C. A comparison of botulinum toxin a and intralesional steroids for the treatment of plantar fasciitis: a randomized, double-blinded study. Foot Ankle Int. 2013 Jan;34(1):8-14. doi: 10.1177/1071100712460215. PMID 23386757
- [Background] Lee WC, Wong WY, Kung E, Leung AK. Effectiveness of adjustable dorsiflexion night splint in combination with accommodative foot orthosis on plantar fasciitis. J Rehabil Res Dev. 2012;49(10):1557-64. doi: 10.1682/jrrd.2011.09.0181. PMID 23516059
- [Background] Probe RA, Baca M, Adams R, Preece C. Night splint treatment for plantar fasciitis. A prospective randomized study. Clin Orthop Relat Res. 1999 Nov;(368):190-5. PMID 10613168
- [Background] Schneider HP, Baca JM, Carpenter BB, Dayton PD, Fleischer AE, Sachs BD. American College of Foot and Ankle Surgeons Clinical Consensus Statement: Diagnosis and Treatment of Adult Acquired Infracalcaneal Heel Pain. J Foot Ankle Surg. 2018 Mar-Apr;57(2):370-381. doi: 10.1053/j.jfas.2017.10.018. Epub 2017 Dec 25. PMID 29284574
- [Background] He C, Ma H. Effectiveness of trigger point dry needling for plantar heel pain: a meta-analysis of seven randomized controlled trials. J Pain Res. 2017 Aug 18;10:1933-1942. doi: 10.2147/JPR.S141607. eCollection 2017. PMID 28860848
- [Background] van de Water AT, Speksnijder CM. Efficacy of taping for the treatment of plantar fasciosis: a systematic review of controlled trials. J Am Podiatr Med Assoc. 2010 Jan-Feb;100(1):41-51. doi: 10.7547/1000041. PMID 20093544
- [Background] Whittaker GA, Munteanu SE, Menz HB, Tan JM, Rabusin CL, Landorf KB. Foot orthoses for plantar heel pain: a systematic review and meta-analysis. Br J Sports Med. 2018 Mar;52(5):322-328. doi: 10.1136/bjsports-2016-097355. Epub 2017 Sep 21. PMID 28935689
- [Background] Diaz Lopez AM, Guzman Carrasco P. [Effectiveness of different physical therapy in conservative treatment of plantar fasciitis: systematic review]. Rev Esp Salud Publica. 2014 Jan-Feb;88(1):157-78. doi: 10.4321/S1135-57272014000100010. Spanish. PMID 24728397
- [Background] Acosta-Olivo C, Simental-Mendia LE, Vilchez-Cavazos F, Pena-Martinez VM, Elizondo-Rodiguez J, Simental-Mendia M. Clinical Efficacy of Botulinum Toxin in the Treatment of Plantar Fasciitis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2022 Feb;103(2):364-371.e2. doi: 10.1016/j.apmr.2021.10.003. Epub 2021 Oct 22. PMID 34688605
- [Background] Buchanan BK, Sina RE, Kushner D. Plantar Fasciitis. 2024 Jan 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK431073/ PMID 28613727
- [Background] Rhim HC, Kwon J, Park J, Borg-Stein J, Tenforde AS. A Systematic Review of Systematic Reviews on the Epidemiology, Evaluation, and Treatment of Plantar Fasciitis. Life (Basel). 2021 Nov 24;11(12):1287. doi: 10.3390/life11121287. PMID 34947818
- [Background] Ahadi T, Nik SS, Forogh B, Madani SP, Raissi GR. Comparison of the Effect of Ultrasound-Guided Injection of Botulinum Toxin Type A and Corticosteroid in the Treatment of Chronic Plantar Fasciitis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Aug 1;101(8):733-737. doi: 10.1097/PHM.0000000000001900. Epub 2021 Oct 8. PMID 34620739
- [Background] Ruiz-Hernandez IM, Gasco-Adrien J, Buen-Ruiz C, Perello-Moreno L, Tornero-Prieto C, Barrantes-Delgado G, Garcia-Gutierrez M, Rapariz-Gonzalez JM, Tejada-Gavela S. Botulinum toxin A versus platelet rich plasma ultrasound-guided injection in the treatment of plantar fasciitis: A randomised controlled trial. Foot Ankle Surg. 2024 Feb;30(2):117-122. doi: 10.1016/j.fas.2023.10.004. Epub 2023 Oct 14. PMID 37949704
- [Background] Hamstra-Wright KL, Huxel Bliven KC, Bay RC, Aydemir B. Risk Factors for Plantar Fasciitis in Physically Active Individuals: A Systematic Review and Meta-analysis. Sports Health. 2021 May-Jun;13(3):296-303. doi: 10.1177/1941738120970976. Epub 2021 Feb 3. PMID 33530860

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT06788158/Prot_SAP_ICF_000.pdf